CLINICAL TRIAL: NCT03615391
Title: Predictive Role and HuR Mechanisms of Regulation in the Brain Tumours
Acronym: HUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/APJC/HUR/GAUCHOTTE/MS
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Brain Tumours
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The HuR protein binds to AU-rich elements in the untranslated 3' region of messenger RNA, thus allowing their stabilization. Its targets include multiple cell cycle regulating proteins, cytokines and growth factors. In some cancers, its overall expression level but especially its cytoplasmic expression are correlated to a higher grade and constitute a poor prognostic factor. To date, HuR's deregulation mechanisms remain poorly understood. A few experimental studies have shown the role of certain microARNS, or of post-translational modifications. In brain tumours, HuR expression, its prognostic value and its deregulation mechanisms have been little studied to date.

The first part of the project will be a monocentric retrospective study of human brain tumour samples collected during biopsies or surgical removal. We will first evaluate HuR expression in 140 brain tumors, including 40 meningiomas and 100 gliomas of increasing grade, and look for a correlation with histological grade and survival. We will then apprehend the consequences of its deregulation by analyzing different factors involved in the cell cycle and stress response markers. Finally, we will study the mechanisms of HuR deregulation by analyzing the expression level of several microRNAs (miR16, miR519) and the methylation state of HuR.

The second part of the project will focus on cell lines from human brain tumours. We will first attempt to confirm the interactions between HuR and markers involved in the cell cycle and stress response, then the regulation of HuR by its methylation and by microRNAs (miR16 and miR519). We would also like to study the consequences of HuR inhibition and overexpression on cell proliferation, under various conditions of induced stress (pharmacological agents, physical stress). Finally, we will study the consequences of an experimental vitamin B12 deficiency on HuR expression and tumor cell adaptation to stress.

ELIGIBILITY:
Inclusion Criteria

* Grade I and II meningiomas (WHO)
* Diffuse grade II glioma (astrocytoma, oligodendroglioma)
* Grade III anaplastic gliomas (astrocytomas and anaplastic oligodendrogliomas)
* Grade IV glioblastoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with braim tumor (meningioma, glioma, glioblastoma)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2012-10-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
level HuR's immunohistochemical expression | at diagnosis
time progression-free | through study completion, an average 3 years
time overall survival | through study completion, an average 3 years

SECONDARY OUTCOMES:
methyl-HuR level | 1 day at diagnosis
PHH3 level | 1 day at diagnosis
MCM6 level | 1 day at diagnosis
Ki-67 level | 1 day at diagnosis
cyclin D1 level | 1 day at diagnosis
Bcl-2 | 1 day at diagnosis
pPERK level | 1 day at diagnosis
ATF6 level | 1 day at diagnosis
SIRT1 level | 1 day at diagnosis
IRE-1α level | 1 day at diagnosis
HIF-1α level | 1 day at diagnosis
caspase 3 activated level | 1 day at diagnosis
VEGF level | 1 day at diagnosis
CARM1 level | 1 day at diagnosis
  Vitamin B12 metabolism
miR16 expression level by qRT-PCR | 1 day at diagnosis
miR519 expression level by qRT-PCR | 1 day at diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Guillaume GAUCHOTTE, Vandœuvre-lès-Nancy, France